CLINICAL TRIAL: NCT01046799
Title: Prevention of HBV Reinfection After Liver Transplantation Using Entecavir Monotherapy After Short-term HBIg Administration: A Pilot Study
Brief Title: Prevention of Hepatitis B Virus Reinfection After Liver Transplantation With Entecavir
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HepNet Study House, German Liverfoundation (Network)
Collaborators: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-005976-28
Record Dates: First submitted 2010-01-09; First posted 2010-01-12 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Liver Transplantation; Hepatitis B; Liver Disease
Keywords: hepatitis B; liver transplantation; shortterm HBIg; lamivudine resistance
MeSH Terms: conditions — Hepatitis B; Liver Diseases | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Entecavir (Experimental)
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — Entecavir monotherapy after short-term HBIg therapy for patients transplanted for hepatitis B induced end-stage liver disease; in case of prior lamivudine treatment, tenofovir will be added to the reinfection prophylaxis
  Other Names: Baraclude

SUMMARY:
The purpose of this study is to determine whether hepatitis B immunoglobin can be discontinued early after hepatitis B virus (HBV) induced liver transplantation and be replaced by the nucleoside analogue entecavir to prevent hepatitis B reinfection.

ELIGIBILITY:
Inclusion Criteria:

* liver transplantation for hepatitis B induced endstage liver disease
* absence of coinfection with HIV and HCV
* female and male patients >= 18 years of age

Exclusion Criteria:

* any evidence of other causes for endstage liver disease
* patients that do not fulfill the criteria for liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-03; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
prevention of hepatitis B virus reinfection one year after liver transplantation with entecavir monotherapy | one year

SECONDARY OUTCOMES:
hepatitis Bs antigen negativity can be maintained by entecavir in the second year after HBV induced liver transplantation | two years

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Manns, MD, Principal Investigator — Hannover Medical School; Heiner Wedemeyer, MD, Principal Investigator — Hannover Medical School
Locations (3):
- Germany (3):
  - University Clinic Essen, Essen
  - Hannover Medical School, Hanover
  - University Hospital Heidelberg, Heidelberg